CLINICAL TRIAL: NCT04324216
Title: Effectiveness of a Combination of Three-dimensional Virtual Reality and Hands-on Aromatherapy in Improving Institutionalized Older Adults' Psychological Health
Brief Title: Three-dimensional Virtual Reality and Hands-on Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201903HM012
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Mental Health
Keywords: 3D VR; Aromatherapy; older adult; happiness; stress; sleep quality; experience on meditation; life satisfaction
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 3D virtual reality and hands-on aromatherapy
  Interventions: Other: 3D virtual reality and hands-on aromatherapy
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: 3D virtual reality and hands-on aromatherapy — Participants will receive 8-session 3DVR aroma therapy activities. Each session was delivered over 2 hours once a week, and at each session, the participant received hands-on guidance for preparing an aromatherapy product that they could use for the next seven days.
  Arms: Experimental group

SUMMARY:
A quasi-experimental trial was designed to evaluate the effectiveness of this combination in promoting happiness, perceived stress, sleep quality, experience on meditation, and life satisfaction among institutionalized older adults in Taiwan.

DETAILED DESCRIPTION:
Background: In Taiwan, which has one of the most rapidly aging populations in the world, it is becoming increasingly critical to promote successful aging strategies that are effective, easily usable, and acceptable to institutionalized older adults. Although many practitioners and professionals have explored aromatherapy and identified its positive psychological benefits, the effectiveness of a combination of 3D virtual reality and hands-on aromatherapy remains unknown.

Objectives: A quasi-experimental trial was designed to evaluate the effectiveness of this combination in promoting happiness, perceived stress, sleep quality, experience on meditation, and life satisfaction among institutionalized older adults in Taiwan.

Methods: Sixty institutionalized elderly participants underwent the combination program or were in a control group. Weekly two-hour sessions were implemented for 9 weeks. The outcome variables were happiness perceived, stress, sleep quality, experience on meditation, and life satisfaction, which were assessed at baseline, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* An ability to understand verbal instructions
* An ability to provide simple responses
* An ability to operate a joystick freely with at least one hand

Exclusion Criteria:

* A history of severe psychiatric conditions;
* Dementia
* Significant visual or hearing impairment;
* Marked upper motor difficulties that could affect the participants' ability to participate in the study
* Currently suffering from severe illnesses, e.g., stroke and Parkinson disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Happiness | nine weeks
  The Oxford Happiness Inventory (OHI) was used to measure happiness. The OHI consists of 29 items, Each item was scored on a Likert-type scale of 1-4, with higher scores indicating a higher level of happiness.
Perceived stress | nine week
  The Perceived Stress Scale (PSS-14) consists of 14 items. Each item was scored on a Likert-type scale that ranged from 0 (never) to four (very often). With higher scores indicating a higher level of stress.
Sleep quality | nine weeks
  The Pittsburgh sleep quality index (PSQI) was consists of 14 items. Each item was scored on a Likert-type scale that ranged from 1 to 4, with higher scores indicating a lower level of sleep quality.
Experience on meditation | nine weeks
  A shortened version of the 10-item Experience on meditation (EOM-EL). Each item was scored on a Likert-type scale of 1-5, with higher scores indicating a higher level of experience on meditation.
Life satisfaction | nine weeks
  This scale is a short-form version containing 10 items from the 20-item Life Satisfaction Index A (LSIA). The response options for scoring were 0 indicating "Disagree" and 1 indicating "Agree". The total raw scores ranged from 0 to 10, with higher scores indicating a higher level of life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai YF, Wong TK, Ku YC. Self-care management of sleep disturbances and risk factors for poor sleep among older residents of Taiwanese nursing homes. J Clin Nurs. 2008 May;17(9):1219-26. doi: 10.1111/j.1365-2702.2007.02020.x. Epub 2008 Feb 11. PMID 18266847
- [Background] Gueldner SH, Loeb S, Morris D, Penrod J, Bramlett M, Johnston L, Schlotzhauer P. A comparison of life satisfaction and mood in nursing home residents and community-dwelling elders. Arch Psychiatr Nurs. 2001 Oct;15(5):232-40. doi: 10.1053/apnu.2001.27020. PMID 11584352
- [Background] Lehrner J, Marwinski G, Lehr S, Johren P, Deecke L. Ambient odors of orange and lavender reduce anxiety and improve mood in a dental office. Physiol Behav. 2005 Sep 15;86(1-2):92-5. doi: 10.1016/j.physbeh.2005.06.031. PMID 16095639
- [Background] Snow LA, Hovanec L, Brandt J. A controlled trial of aromatherapy for agitation in nursing home patients with dementia. J Altern Complement Med. 2004 Jun;10(3):431-7. doi: 10.1089/1075553041323696. PMID 15253846
- [Background] Kim S, Song JA, Kim ME, Hur MH. [Effects of Aromatherapy on Menopausal Symptoms, Perceived Stress and Depression in Middle-aged Women: A Systematic Review]. J Korean Acad Nurs. 2016 Oct;46(5):619-629. doi: 10.4040/jkan.2016.46.5.619. Korean. PMID 27857006
- [Background] Tang SK, Tse MY. Aromatherapy: does it help to relieve pain, depression, anxiety, and stress in community-dwelling older persons? Biomed Res Int. 2014;2014:430195. doi: 10.1155/2014/430195. Epub 2014 Jul 13. PMID 25114901
- [Background] Kim ME, Jun JH, Hur MH. [Effects of Aromatherapy on Sleep Quality: A Systematic Review and Meta-Analysis]. J Korean Acad Nurs. 2019 Dec;49(6):655-676. doi: 10.4040/jkan.2019.49.6.655. Korean. PMID 31932562
- [Background] Redstone L. Mindfulness meditation and aromatherapy to reduce stress and anxiety. Arch Psychiatr Nurs. 2015 Jun;29(3):192-3. doi: 10.1016/j.apnu.2015.03.001. Epub 2015 Mar 13. No abstract available. PMID 26001720
- [Background] Lua PL, Salihah N, Mazlan N. Effects of inhaled ginger aromatherapy on chemotherapy-induced nausea and vomiting and health-related quality of life in women with breast cancer. Complement Ther Med. 2015 Jun;23(3):396-404. doi: 10.1016/j.ctim.2015.03.009. Epub 2015 Apr 21. PMID 26051575
- [Background] Hsu MC, Creedy D, Moyle W, Venturato L, Tsay SL, Ouyang WC. Use of Complementary and Alternative Medicine among adult patients for depression in Taiwan. J Affect Disord. 2008 Dec;111(2-3):360-5. doi: 10.1016/j.jad.2008.03.010. Epub 2008 Apr 28. PMID 18442859
- [Background] Yang YP, Lee FP, Chao HC, Hsu FY, Wang JJ. Comparing the Effects of Cognitive Stimulation, Reminiscence, and Aroma-Massage on Agitation and Depressive Mood in People With Dementia. J Am Med Dir Assoc. 2016 Aug 1;17(8):719-24. doi: 10.1016/j.jamda.2016.03.021. Epub 2016 May 7. PMID 27168052
- [Background] Hwang E, Shin S. The effects of aromatherapy on sleep improvement: a systematic literature review and meta-analysis. J Altern Complement Med. 2015 Feb;21(2):61-8. doi: 10.1089/acm.2014.0113. Epub 2015 Jan 13. PMID 25584799
- [Background] Babakhanian M, Ghazanfarpour M, Kargarfard L, Roozbeh N, Darvish L, Khadivzadeh T, Dizavandi FR. Effect of Aromatherapy on the Treatment of Psychological Symptoms in Postmenopausal and Elderly Women: A Systematic Review and Meta-analysis. J Menopausal Med. 2018 Aug;24(2):127-132. doi: 10.6118/jmm.2018.24.2.127. Epub 2018 Aug 31. PMID 30202763
- [Background] Chang SY. [Effects of aroma hand massage on pain, state anxiety and depression in hospice patients with terminal cancer]. Taehan Kanho Hakhoe Chi. 2008 Aug;38(4):493-502. doi: 10.4040/jkan.2008.38.4.493. Korean. PMID 18753801
- [Background] Wilkinson SM, Love SB, Westcombe AM, Gambles MA, Burgess CC, Cargill A, Young T, Maher EJ, Ramirez AJ. Effectiveness of aromatherapy massage in the management of anxiety and depression in patients with cancer: a multicenter randomized controlled trial. J Clin Oncol. 2007 Feb 10;25(5):532-9. doi: 10.1200/JCO.2006.08.9987. PMID 17290062
- [Background] Tiran D, Chummun H. Complementary therapies to reduce physiological stress in pregnancy. Complement Ther Nurs Midwifery. 2004 Aug;10(3):162-7. doi: 10.1016/j.ctnm.2004.03.006. PMID 15279857
- [Background] Atsumi T, Tonosaki K. Smelling lavender and rosemary increases free radical scavenging activity and decreases cortisol level in saliva. Psychiatry Res. 2007 Feb 28;150(1):89-96. doi: 10.1016/j.psychres.2005.12.012. Epub 2007 Feb 7. PMID 17291597
- [Background] Smith MC, Kyle L. Holistic foundations of aromatherapy for nursing. Holist Nurs Pract. 2008 Jan-Feb;22(1):3-9; quiz 10-1. doi: 10.1097/01.HNP.0000306321.03590.32. PMID 18172401
- [Background] Sayorwan W, Siripornpanich V, Piriyapunyaporn T, Hongratanaworakit T, Kotchabhakdi N, Ruangrungsi N. The effects of lavender oil inhalation on emotional states, autonomic nervous system, and brain electrical activity. J Med Assoc Thai. 2012 Apr;95(4):598-606. PMID 22612017
- [Background] Bouya S, Ahmadidarehsima S, Badakhsh M, Balouchi A, Koochakzai M. Effect of aromatherapy interventions on hemodialysis complications: A systematic review. Complement Ther Clin Pract. 2018 Aug;32:130-138. doi: 10.1016/j.ctcp.2018.06.008. Epub 2018 Jun 13. PMID 30057040
- [Background] Kim MJ, Nam ES, Paik SI. [The effects of aromatherapy on pain, depression, and life satisfaction of arthritis patients]. Taehan Kanho Hakhoe Chi. 2005 Feb;35(1):186-94. doi: 10.4040/jkan.2005.35.1.186. Korean. PMID 15778570
- [Background] Soden K, Vincent K, Craske S, Lucas C, Ashley S. A randomized controlled trial of aromatherapy massage in a hospice setting. Palliat Med. 2004 Mar;18(2):87-92. doi: 10.1191/0269216304pm874oa. PMID 15046404
- [Background] Shin ES, Seo KH, Lee SH, Jang JE, Jung YM, Kim MJ, Yeon JY. Massage with or without aromatherapy for symptom relief in people with cancer. Cochrane Database Syst Rev. 2016 Jun 3;2016(6):CD009873. doi: 10.1002/14651858.CD009873.pub3. PMID 27258432
- [Derived] Cheng VY, Huang CM, Liao JY, Hsu HP, Wang SW, Huang SF, Guo JL. Combination of 3-Dimensional Virtual Reality and Hands-On Aromatherapy in Improving Institutionalized Older Adults' Psychological Health: Quasi-Experimental Study. J Med Internet Res. 2020 Jul 23;22(7):e17096. doi: 10.2196/17096. PMID 32706660